CLINICAL TRIAL: NCT04861493
Title: Cathelicidin LL-37 Levels in the Gingival Crevicular Fluid and the Saliva of Smokers and Non-smokers With Stage III,IV Periodontitis :An Observational Study
Brief Title: Cathelicidin LL-37 Levels in the GCF and the Saliva of Smokers and Non-smokers With Stage III,IV Periodontitis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Magdy Abu El Eneen, principle investigator, Cairo University
Other Study IDs: 9221
Record Dates: First submitted 2021-04-18; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Smoking Reduction
MeSH Terms: conditions — Smoking Reduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid samples Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Smokers with stage III,IV periodontitis: patients with stage III,IV periodontitis having CAL>5 mm and PD>5 mm in one or more sites and bleeding on probing >30% and smoking at least 10 cigarettes /day for a minmum of 5 years.
- Non-smokers with stage III,IV periodontitis: patients with stage III,IV periodontitis having CAL>5 mm and PD>5 mm in one or more sites and bleeding on probing >30% and they are never smoked before.
- Healthy patients: patients free from periodontitis or any systemic disease and never smoked before.

SUMMARY:
Periodontitis is considered an inflammatory disease that results in the disruption of oral hemeostasis and is associated with the presence of dental plaque influenced by genetic and environmental factors. It is well-establised that smokers have an increased severity of periodontal disease,a higher prevalance of tooth loss and total edentulism.

DETAILED DESCRIPTION:
Antimicrobial peptides (AMPs) are soluble molecules participating in the innate immunity of mucosal surfaces against pathogens. Dysregulated expression of AMPs has been considered a possible causal mechanistic link in the microbial dysbiosis associated with periodontal disease and some risk factors, including tobacco smoking, diabetes mellitus, and obesity.Antimicrobial peptides as a part of innate immunity are important molecules that provide a balance between disease and health. Moreover, they are considered to be an important intermediate step in initiating an initial immune response against the microbial side of the gingival epithelium and in the transition to acquired immunity. Cathelicidins, in particular - which play an important role in regulating the immunological response of oral tissues, are a group of peptides released from neutrophil granules and they are present only in humans in the form of LL-37.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a minimum of 15 natural teeth.
2. At least four non-adjacent teeth sites in each jaw having CAL ≥ 5 mm and PD > 5 mm in one or more sites.
3. Bleeding on probing (BOP) ≥ 30%.
4. Tooth loss due to periodontitis ≤ 4 teeth.
5. For smoker's patients; study will include patients who regularly smoked at least 10 cigarettes/day for a minimum of 5 years.
6. For non-smokers patients; study will include patients who had never smoked.

Exclusion Criteria:

1. Individuals with a history of systemic diseases or immunological disorders.
2. Individuals using hormone replacement therapy.
3. Pregnant and lactating women.
4. Individuals that received periodontal treatment within the last 6 months.
5. Individuals with a history of systemic antibiotics and anti-inflammatory drugs within the last 3 months.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Group 1: Smokers with stage III,IV periodontitis Group 2: Non-smokers with stage III,IV periodontitis Group 3: Healthy patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
LL-37 levels in the GCF and saliva | Through study completion,an average of 1 year
  GCF,Saiva sampling to assess LL-37 levels by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Ghallab, Study Director — main supervisor
Locations (1):
- Faculty of dentistry cairo university, Al Manyal, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes